CLINICAL TRIAL: NCT01135745
Title: Reclaim® Deep Brain Stimulation Therapy for Obsessive-Compulsive Disorder: Post-Market Clinical Follow-up Study (OCD PMCF)
Brief Title: Deep Brain Stimulation for Obsessive Compulsive Disorder (OCD PMCF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCD PMCF Study 1.02.7003
Record Dates: First submitted 2010-05-05; First posted 2010-06-03 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deep Brain Stimulation Therapy for OCD (Experimental): Reclaim® DBS Therapy uses thin wires to deliver electric current (stimulation) to a very specific target in the brain. These wires are implanted surgically. They are attached to internal neurostimulators implanted under the skin of the chest below the collarbone, similar to cardiac pacemakers, or in the abdominal wall. The study doctor will adjust the settings of the electrical stimulation to optimize treatment for each participant.
  Interventions: Device: Reclaim® Deep Brain Stimulation

INTERVENTIONS:
Device: Reclaim® Deep Brain Stimulation — Implant of leads in pre-defined brain area; implant of neurostimulators

SUMMARY:
The purpose of the study is to monitor the safety and performance of Reclaim® Deep Brain Stimulation (DBS) Therapy in patients with chronic, severe, treatment-resistant Obsessive Compulsive Disorder.

DETAILED DESCRIPTION:
OCD is an anxiety disorder characterized by intrusive thoughts or images (obsessions), which increase anxiety, commonly accompanied by repetitive or ritualistic actions (compulsions), which decrease anxiety. The most frequent symptoms are contamination concerns with consequent washing or concerns about harm to self or others with consequent checking.

Although many OCD patients benefit from pharmacotherapy or CBT, between 7% and 10% of OCD patients fail to benefit from these standard treatments and may be considered treatment-resistant with a chronic deteriorating course. The most severely afflicted and disabled of these patients may be indicated for neurosurgical treatments, often considered as a therapy of last resort.

Neurosurgical procedures currently used in the treatment of severe, treatment-resistant OCD include anterior cingulotomy, subcaudate tractotomy, limbic leucotomy (which is a combination of the first two procedures) and anterior capsulotomy. The commonality between the different neurosurgical procedures is the irreversible lesioning of bilateral neuroanatomical structures and/or interconnecting pathways that are believed to be involved in the control of affect and limbic function.

An alternative neurosurgical treatment option to the standard lesioning procedures is Reclaim® Deep Brain Stimulation (DBS) Therapy for OCD, which received CE mark in July 2009.

ELIGIBILITY:
Inclusion Criteria:

* signing and dating of Informed Consent
* male and female patients at least 18 years of age
* diagnosis of Obsessive Compulsive Disorder
* meeting the definition of treatment resistance

Exclusion Criteria:

* Axis-I disorder primary to OCD
* contraindication to implantation
* suicide risk
* risk of non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Characterization of Adverse Events related to implant procedures, device or stimulation | 12 months
  Prior to any other study procedures Adverse Events will be assessed at every study visit, i.e. after assessment at the baseline visit this will be implant visit, first parameter selection visit and regular visits after 3, 6, and 12 months treatment. AEs will also be collected at all unscheduled visits prior to all other assessments. AEs and stimulation effects will be categorized and recorded in the patient CRF. An independent clinical event committee will review and adjudicate AEs on a regular basis throughout the study.

SECONDARY OUTCOMES:
To characterize improvement from baseline in OCD symptoms assessed by YBOCS. | 12 months
  YBOCS score is taken at baseline and then at post-implant visits after 3, 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Loes Gabriels, MD PhD MsEng, Principal Investigator — Professor of Psychiatry at UZ Leuven; Andreas Wahl-Kordon, MD, Principal Investigator — University Hospital Lübeck; Ludger Tebartz van Elst, MD, Principal Investigator — University Hospital Freiburg; Jose M Menchon, MD, Principal Investigator — University Hospital Bellvitge Barcelona; Antonio Higueras, MD, Principal Investigator — University Hospital Granada; Orsola Gambini, MD, Principal Investigator — University Hospital San Paolo Milan; Michael Schüpbach, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern; Siegried Kasper, MD, Principal Investigator — Department of Psychiatry and Psychotherapy Medical University of Vienna; Diana Radu-Djurfeldt, Principal Investigator — Karolinska Institutet, Stockholm; Renana Eitan, Principal Investigator — Hadassah-Hebrew University and Medical Center, Jerusalem
Locations (8):
- Universitaire Ziekenhuis Leuven, Leuven, Belgium
- Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck, Germany
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel
- A.O. San Paolo Polo Universitario, Milan, Italy
- Spain (2):
  - Hospital Ciutat Sanitaria I Universitaria de Bellvitge, Barcelona
  - Hospital Virgen de las Nieves, Granada
- Karolinska University Hospita, Stockholm, Sweden
- Inselspital Bern, Bern, Switzerland

REFERENCES:
- [Background] Rauch SL, Dougherty DD, Malone D, Rezai A, Friehs G, Fischman AJ, Alpert NM, Haber SN, Stypulkowski PH, Rise MT, Rasmussen SA, Greenberg BD. A functional neuroimaging investigation of deep brain stimulation in patients with obsessive-compulsive disorder. J Neurosurg. 2006 Apr;104(4):558-65. doi: 10.3171/jns.2006.104.4.558. PMID 16619660